CLINICAL TRIAL: NCT03081663
Title: Cost and Patient Satisfaction After Total Knee Arthroplasty: Standard Medial Para-patellar Versus Quadriceps Sparing Mid-vastus Surgical Approach
Brief Title: Quadriceps Sparing Versus Standard Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Brent Lanting, Orthopaedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 108949
Record Dates: First submitted 2017-03-08; First posted 2017-03-16 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis; Knee Arthroplasty
Keywords: total knee arthroplasty; quadriceps sparing mid-vastus; medial para-patellar
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to undergo their surgery through either the quadriceps-sparing mid-vastus approach or the medial para-patellar approach and with or without a tourniquet. We will stratify based on which type of analgesia will be used post-surgery, either an adductor canal block or local infiltration.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be told which group they have been assigned to until they have reached the final follow-up visit for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Quads-Sparing Approach with Tourniquet (Experimental): Participants will have a navigated total knee arthroplasty with a quadriceps-sparing mid-vastus approach and a tourniquet.
  Interventions: Procedure: Quads-Sparing Approach
- Medial Para-Patellar with Tourniquet (Active Comparator): Participants will undergo total knee arthroplasty with a medial para-patellar approach and a tourniquet. An intramedullary femoral guide and extramedullary tibial guide will be used during the surgery.
  Interventions: Procedure: Medial Para-Patellar Approach
- Quads-Sparing Approach w/o Tourniquet (Active Comparator): Participants will have a navigated total knee arthroplasty with a quadriceps-sparing mid-vastus approach and no tourniquet.
  Interventions: Procedure: Quads-Sparing Approach
- Medial Para-Patellar w/o Tourniquet (Active Comparator): Participants will undergo total knee arthroplasty with a medial para-patellar approach and no tourniquet. An intramedullary femoral guide and extramedullary tibial guide will be used during the surgery.
  Interventions: Procedure: Medial Para-Patellar Approach

INTERVENTIONS:
Procedure: Quads-Sparing Approach — Quadriceps-sparing mid-vastus approach for total knee arthroplasty
  Other Names: quads-sparing
  Arms: Quads-Sparing Approach w/o Tourniquet; Quads-Sparing Approach with Tourniquet
Procedure: Medial Para-Patellar Approach — Medial para-patellar approach for total knee arthroplasty
  Other Names: standard
  Arms: Medial Para-Patellar w/o Tourniquet; Medial Para-Patellar with Tourniquet

SUMMARY:
This study is a randomized clinical trial comparing standard medial para-patellar total knee arthroplasty with a quadriceps sparing mid-vastus approach. Patients who are medically well and have a good support structure at home will be randomized to a standard or quadriceps sparing surgical approach stratified by type of analgesia (adductor canal block or local infiltration). We will compare patient satisfaction and costs from the perspective of the Ministry of Health, the institution, society and the patient.

DETAILED DESCRIPTION:
Over the past 20 years the length of stay in hospital after total knee replacements has decreased from 9 days to 3 days in Canada and in just the last 10 years the mean length of stay has decreased by half from 6 to 3 days. In order to discharge patients quicker from hospital it's been theorized that less invasive techniques and better, longer lasting anaesthesia are required.

The less invasive quadriceps sparing mid-vastus approach for TKA has been compared to the standard medial para-patellar technique in many studies. Meta-analyses that have looked at studies comparing these approaches have shown some early advantages for quadriceps sparing early post-surgery, but no differences between groups later on and no difference in complications. Early advantages of the mid-vastus approach could potentially allow for earlier and safer discharge from hospital.

Adductor canal block (ACB) and local infiltration analgesia (LIA) form the mainstay of opioid sparing multimodal analgesia for TKA. The nerves of the adductor canal innervate the superficial and deep tissues of the anterior and medial aspects of the knee. ACB has been shown to provide equivalent analgesia while maintaining quadriceps power compared to femoral nerve block (FNB). LIA involves infiltrating the soft tissues of the posterior, lateral and medial aspects of the knee with local anesthetics, ketorolac and morphine. Due to their minimal impact on motor function, ACB and LIA are suitable for fast track TKA.

In combination, quadriceps sparing mid-vastus TKA with ACB may allow patients to be discharged from hospital quicker when compared with standard medial para-patellar TKA with LIA. With our study we aim to investigate whether a quadriceps sparing TKA can provide cost savings without changing complication rates when compared to the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* patients requiring primary total knee replacement
* patients willing and able to comply with follow-up requirements and self-evaluations
* patients willing to sign an IRB approved informed consent form
* English fluency (printed instructions are provided in English only)
* varus arthropathy
* osteoarthritis
* ASA less than or equal to 3
* home/cell phone access
* adult to accompany patient home post-operatively and to stay with patient for a minimum period of 1-2 days

Exclusion Criteria:

* patients with inflammatory arthritis
* patients with a BMI greater than 40 or less than 18
* patients who are skeletally immature
* patient with an active infection or suspected latent infection in or about the joint
* bone stock that is inadequate for support or fixation of the prosthesis
* hardware precluding intramedullary instrumentation
* prior osteotomies of the femur or tibia
* patients living greater than 1.5 hours from the hospital
* patients without access to caregivers, or unable to go to their home after surgery
* cognitive or neuromotor conditions
* patient has significant pain management issues
* patient/family history of anaesthesia related complications (e.g. malignant hypothermia, pseudocholinesterase deficiency, airway difficulties, obstructive sleep apnea)
* significant psycho/social issues that would prevent the patient from managing at home safely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
Indirect and Direct Costs of Treatment | 1 year
  ER visits, clinician visits, caregiver lost productivity, tests, etc.

SECONDARY OUTCOMES:
Pain Numeric Rating Scale | 1 year
  Pain
Short Form - 12 (SF-12) | 1 year
  Quality of Life
Western Ontario McMaster Osteoarthritis Index (WOMAC) | 1 year
  Functional Outcome
Knee Society Score (KSS) | 1 year
  Functional Outcome
EuroQol-5D (EQ-5D) | 1 year
  Quality of Life
Timed Up and Go Test | 1 year
  Function
Adverse events | 1 year
  Falls, wound problems, pulmonary embolism, deep vein thrombosis, infection, etc.
Caregiver Assistance Scale | 6 weeks
  Caregiver Confidence
Caregiver Strain Index | 6 weeks
  Caregiver Strain
Patient Satisfaction Questionnaire | 2 weeks
  Patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Lanting, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No